CLINICAL TRIAL: NCT01793870
Title: A Four Way Crossover Study in Healthy Volunteers to Evaluate the Application of Stable Isotope Approach to Reduce Number of Subjects Needed for PK Studies
Brief Title: A Study in Healthy Volunteers to Evaluate the Application of Stable Isotope Approach to Reduce Number of Subjects Needed for PK Studies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 117058
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Metabolic, Cardiovascular
Keywords: pharmacokinetic; carvedilol; Stable isotope technique
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (27.5 mg total maximum dose) (Experimental): Single oral dose of carvedilol (25 milligram [mg]) as a 1 x 25 mg immediate release tablet and up to 2.5 mg of enriched carvedilol drug substance under fasted conditions.
  Interventions: Drug: Tab carvedilol 25 mg; Drug: Powder carvedilol up to 2.5 mg
- Treatment B (27.5 mg total maximum dose) (Experimental): Single oral dose of carvedilol (25 mg) as a 1 x 25 mg immediate release tablet and up to 2.5 mg of enriched carvedilol drug substance under fasted conditions.
  Interventions: Drug: Tab carvedilol 25 mg; Drug: Powder carvedilol up to 2.5 mg
- Treatment C (33.75 mg total maximum dose) (Experimental): Single oral dose of carvedilol (31.25 mg) as a 1 x 25 mg immediate release tablet, a 1 x 6.25 mg immediate release tablet and up to 2.5 mg of enriched carvedilol drug substance under fasted conditions.
  Interventions: Drug: Tab carvedilol 25 mg; Drug: Tab carvedilol 6.25 mg; Drug: Powder carvedilol up to 2.5 mg
- Treatment D (27.5 mg total maximum dose) (Experimental): Single oral dose of carvedilol (25 mg) as a 1 x 25 mg x immediate release tablet and up to 2.5 mg of enriched carvedilol drug substance under fed conditions.
  Interventions: Drug: Tab carvedilol 25 mg; Drug: Powder carvedilol up to 2.5 mg

INTERVENTIONS:
Drug: Tab carvedilol 25 mg — Carvedilol 25 mg immediate release tablet
Drug: Tab carvedilol 6.25 mg — Carvedilol 6.25 mg immediate release tablet
  Arms: Treatment C (33.75 mg total maximum dose)
Drug: Powder carvedilol up to 2.5 mg — Carvedilol up to 2.5 mg isotopically enriched drug substance powder

SUMMARY:
This will be a randomized, open-label, single dose, 4-period, period balanced, crossover study. There will be at least 5 days between dosing in each session. The study consists of Screening period (30 days prior to Day 1), Treatment period consisting of 4 dosing periods (Day 1 is the dosing day and Day 2) and Follow-up period (7-14 days post-last dose).

The detailed treatment regimen will be A and B (27.5 mg total maximum dose): Single oral dose of carvedilol 25 mg immediate release tablet and up to 2.5 mg of enriched carvedilol powder under fasted conditions; C (33.75 mg total maximum dose): Single oral dose of carvedilol 31.25 mg as 25 mg immediate release tablet, a 6.25 mg immediate release tablet and up to 2.5 mg of enriched carvedilol powder under fasted conditions; D (27.5 mg total maximum dose): Single oral dose of carvedilol 25 mg immediate release tablet and up to 2.5 mg of enriched carvedilol powder under fed conditions. Approximately 15 subjects will be randomized to receive one of four treatment sequences (ADBC, BACD, CBDA, or DCAB).

The pharmacokinetic sampling and safety data will be collected in the Treatment period (Day 1 and 2).

ELIGIBILITY:
Inclusion criteria

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG monitoring.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential Female subjects of child bearing potential must agree to use contraception from screening until the follow-up visit.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods.
* Body weight >= 50 kilogram (kg) and BMI within the range 18.5 to 29.9 kilogram per meter square (kg/m^2) (inclusive).
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Average QT corrected using Bazett's formula (QTcB) or QT corrected using Fridericia's formula (QTcF) <450 milliseconds (msec).
* Suitable for cannulation and with adequate venous access. Exclusion criteria
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Resting heart rate of <50 beats per minute (bpm) at screening
* Any of the following abnormalities on 12-lead electrocardiogram (ECG) during screening: conduction abnormalities denoted by any of the following- PR interval <120 msec or >200 msec; non-specific IVCD (intra-ventricular conduction delay) with QRS duration >=110 msec and where the morphology does NOT meet criteria for left (LBBB) or right bundle branch block (RBBB); incomplete RBBB as defined by QRS duration >=100 msec but <120 msec with RBBB pattern; complete RBBB and LBBB; evidence of second- or third- degree atrio ventricular (AV) block; pathological Q-waves (Q-wave wider than 0.04 sec or depth not greater than 0.4-0.5 millivolt [mV]); evidence of ventricular pre-excitation; evidence of left axis deviation (left axis deviation is -30 to -90 degrees) but not normal leftward axis, ST-T wave abnormalities.
* Documented history of low blood pressure (average systolic blood pressure [SBP] <= 110 millimeters of mercury [mm Hg] and/or DBP <=60 mm Hg) or semi-supine blood pressure below these values at time of screening.
* Orthostatic hypotension diagnosed at screening (orthostatic hypotension will be defined as a reduction in systolic blood pressure of 20 mm Hg or more and/or a reduction in diastolic blood pressure of 10 mmHg or more within three minutes of standing upright from supine at screening).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to adhere with restrictions detailed in the informed consent or protocol.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Subject is a smoker, based on at least 12 months non-smoking history.
* Lactating females.
* Subjects who have asthma or a history of asthma or of bronchospasm. Subjects with a history of childhood asthma but are now asymptomatic may be included at the investigators discretion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2013-06-17 (Actual); Study Completion 2013-06-17 (Actual)

PRIMARY OUTCOMES:
The AUC for both the enriched and non-enriched R- and S-isomers of carvedilol | Day 1:pre-dose, 15 minutes (mins), 30 mins, 45 mins, 1 hour (h), 2 h, 3 h, 4 h, 6 h, 8 h and 12 h post-dose; Day 2: at 24 h and 36 h post dose
  The pharmacokinetic parameters will include area under the time concentration curve (AUC) for both the enriched and non-enriched R- and S-isomers of carvedilol
The Cmax for both the enriched and non-enriched R- and S-isomers of carvedilol | Day 1:pre-dose, 15 minutes (mins), 30 mins, 45 mins, 1 hour (h), 2 h, 3 h, 4 h, 6 h, 8 h and 12 h post-dose; Day 2: at 24 h and 36 h post dose
  The pharmacokinetic parameters will include maximum drug concentration (Cmax) for both the enriched and non-enriched R- and S-isomers of carvedilol

SECONDARY OUTCOMES:
The Tmax for both the enriched and non-enriched R- and S-isomers of carvedilol (as data permit) | Day 1:pre-dose, 15 minutes (mins), 30 mins, 45 mins, 1 hour (h), 2 h, 3 h, 4 h, 6 h, 8 h and 12 h post-dose; Day 2: at 24 h and 36 h post dose
  The pharmacokinetic parameter will include the time when maximum drug concentration is reached (Tmax) for both the enriched and non-enriched R- and S-isomers of carvedilol
The T1/2 for both the enriched and non-enriched R- and S-isomers of carvedilol (as data permit) | Day 1:pre-dose, 15 minutes (mins), 30 mins, 45 mins, 1 hour (h), 2 h, 3 h, 4 h, 6 h, 8 h and 12 h post-dose; Day 2: at 24 h and 36 h post dose
  The pharmacokinetic parameter will include the half life of the drug (T1/2) for both the enriched and non-enriched R- and S-isomers of carvedilol

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 117058 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117058?search=study&study_ids=117058#rs